CLINICAL TRIAL: NCT03804970
Title: Information, Networks and Rewards to Optimise Adherence to Diabetic Services: "INROADS in China": A Randomized Trial
Brief Title: Information, Networks and Rewards to Optimise Adherence to Diabetic Services
Acronym: INROADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Yangxi people hospital, Yangjiang, Guangdong Province (Unknown)
Responsible Party: Principal Investigator, Congdon Nathan, Professor of Preventative Ophthalmology, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ZOC-INROADS
Record Dates: First submitted 2019-01-08; First posted 2019-01-15 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2019-01

CONDITIONS: Diabetes
Keywords: Diabetes; follow-up; Diabetic retinopathy; Diabetic teaching; SMS; rewards
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): Cash rewards for the fellow up+SMS reminders for participants and their family+Showing retinal photos to participants+ Having the Diabetic Club+Watching brief video and basic explanation for disease
  Interventions: Behavioral: cash rewards for the fellow up; Behavioral: Showing retinal photos to participants; Behavioral: SMS reminders for participants and their family; Behavioral: Having the Diabetic Club
- Adjusted intervention group (Experimental): Cash rewards for the fellow up+SMS reminders for participants and their family+Showing retinal photos to participants+Having the Diabetic Club+Watching brief video and basic explanation for disease( But the intensity of intervention based on the severity of diabetic disease)
  Interventions: Behavioral: cash rewards for the fellow up; Behavioral: Showing retinal photos to participants; Behavioral: SMS reminders for participants and their family; Behavioral: Having the Diabetic Club
- Control group (Active Comparator): Watching brief video and basic explanation for disease
  Interventions: Behavioral: Watching brief video and basic explanation for disease

INTERVENTIONS:
Behavioral: cash rewards for the fellow up — This is a multiple stimulus intervention study, and there are two intervention groups. One is the normal intervention group, and the other is the adjusted intervention group. The intensity of intervention in the latter group is based on the severity of diabetic disease.
  Arms: Adjusted intervention group; Intervention group
Behavioral: Showing retinal photos to participants — This is a multiple stimulus intervention study, and there are two intervention groups. One is the normal intervention group, and the other is the adjusted intervention group. The intensity of intervention in the latter group is based on the severity of diabetic disease.
  Arms: Adjusted intervention group; Intervention group
Behavioral: SMS reminders for participants and their family — This is a multiple stimulus intervention study, and there are two intervention groups. One is the normal intervention group, and the other is the adjusted intervention group. The intensity of intervention in the latter group is based on the severity of diabetic disease.
  Arms: Adjusted intervention group; Intervention group
Behavioral: Watching brief video and basic explanation for disease — This basic explanation will be offered by professional doctors or nurses.
  Arms: Control group
Behavioral: Having the Diabetic Club — This is a multiple stimulus intervention study, and there are two intervention groups. One is the normal intervention group, and the other is the adjusted intervention group. The intensity of intervention in the latter group is based on the severity of diabetic disease.
  Arms: Adjusted intervention group; Intervention group

SUMMARY:
This prospective, randomised controlled trial is to investigate whether the complex intervention, including incentives (inexpensive cellphone top-ups), information (viewing one's own fundus photos and receiving SMS informational reminders) and peer support (Diabetes clubs), improve compliance with eye care among rural persons living with diabetes in southern China.

DETAILED DESCRIPTION:
Background: Diabetes affects some 10% of rural-dwellers in southern China. Demand for care of both diabetes and DR is low in this population: Only 25% are in care for diabetes (vs 100% of a matched urban cohort), 0% were being treated for DR (vs 55% of the urban cohort) and 31% said they were likely/very likely to accept diabetic eyecare when it was described to them (vs 78% of the urban group). A simple intervention of informational SMS reminders could significantly increase knowledge about DR and satisfaction with care among rural dwellers, while tripling their compliance with scheduled eye examinations. However, even in the group receiving the SMS reminders, over half failed to present for exams. More effective interventions are needed.

Participants: All the participants with treated diabetes or HbA1c >=6.5% from the Guangdong (Yangjiang) centre of our population-based Rural Diabetic Eye Disease Survey. They must be aged 50-90 years, own a cell phone (ownership is > 95% in the area), have no mobility limitations precluding routine clinic visits or bilateral blindness (<6/120), and be capable of giving informed consent.

Randomisation: To avoid contamination, we are clustering recruitment and randomisation at the level of village and inviting participants in the two study groups to the Yangjiang eye screening centre for follow-up on different clinic days. Block randomization, at village level, will be balanced by the distribution of education levels and travel times from screening centre.

Intervention. All groups will be offered a brief video, already created and piloted, explaining basic information about diabetes and diabetic eye disease. The Intervention group will also receive (i) non-cash rewards (free eye care and modest mobile phone top ups in return for attendance at retinopathy screenings), the value of which will increase with the risk of vision loss (based on existing level of eye disease and HbA1c). (ii) Informational reminders delivered by SMS text 1 day and 1 week prior to scheduled eye exams. In keeping with health economic research,3 the reminders will emphasize anticipated regret: "Your next eye screening visit is next week, on dd/mm/yy. If you miss your eye screening visit, you might regret this if you subsequently lose your vision."; and (iii) peer and village health worker (VHW) networking (supported by the existing Orbis CREST project). Peer supporters will be a nominated family member or friend who has regular contact with the patient and a VHW or a community member with diabetes who has been trained to run monthly group educational sessions in the local village on optimum self-care and self-management of diabetes/DR. An important function of the family member or peer supporter is also to re-inforce the SMS informational reminders before the scheduled clinic visit.

Primary outcome measure: Proportion of scheduled eye care visits attended over 1 year. Secondary outcomes, not the direct target of our intervention, but which might be improved by a behavioural spill-over effect, will include: follow-up HbA1c; medication adherence; retinopathy grade and visual acuity in the better seeing eye.

Power and sample size: Assuming an effect size d= 0.44, and an attrition of 15% over two years, a full trial of 412 patients (42 villages in each of the two groups and 206 patients per group) would have 90% power (two sided alpha error 0.05).

ELIGIBILITY:
Inclusion Criteria:

* They must be aged 50-90 years;
* Own a cell phone (ownership is > 95% in the area);
* Have no mobility limitations precluding routine clinic visits or bilateral blindness (<6/120);
* Be capable of giving informed consent.

Exclusion Criteria:

* Have other serious eye disease;
* Have mobility limitations precluding routine clinic visits or bilateral blindness (<6/120).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Proportion of scheduled eye care visits attended over 1 year | One year
  The visits will be recorded during the 1 year

SECONDARY OUTCOMES:
Follow-up HbA1c | One year
  This outcome will be recorded in the baseline and end-line examination
Proportion of scheduled endocrine care visits attended over 1 year | One year
  The outcome will be recorded during the 1 year
Retinopathy grade in the better seeing eye. | One year
  This outcome will be recorded in the baseline and end-line examination
Visual acuity in the better seeing eye. | One year
  This outcome will be recorded in the baseline and end-line examination

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD, Principal Investigator — Zongshan Ophthalmic Center; Wenyong Huang, MD, Principal Investigator — Zongshan Ophthalmic Center; Chunhui Chen, Study Director — Yangxi People hospital, Guangdong; Congyao Wang, Study Chair — Zongshan Ophthalmic Center
Locations (1):
- Yangxi hospital, Yangjiang, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jin G, Xiao W, Ding X, Xu X, An L, Congdon N, Zhao J, He M. Prevalence of and Risk Factors for Diabetic Retinopathy in a Rural Chinese Population: The Yangxi Eye Study. Invest Ophthalmol Vis Sci. 2018 Oct 1;59(12):5067-5073. doi: 10.1167/iovs.18-24280. PMID 30357401
- [Background] Chen T, Zhu W, Tang B, Jin L, Fu H, Chen Y, Wang C, Zhang G, Wang J, Ye T, Xiao D, Vignarajan J, Xiao B, Kanagasingam Y, Congdon N. A Mobile Phone Informational Reminder to Improve Eye Care Adherence Among Diabetic Patients in Rural China: A Randomized Controlled Trial. Am J Ophthalmol. 2018 Oct;194:54-62. doi: 10.1016/j.ajo.2018.07.006. Epub 2018 Jul 24. PMID 30053472
- [Background] Whitaker KL, Good A, Miles A, Robb K, Wardle J, von Wagner C. Socioeconomic inequalities in colorectal cancer screening uptake: does time perspective play a role? Health Psychol. 2011 Nov;30(6):702-9. doi: 10.1037/a0023941. Epub 2011 May 30. PMID 21639637
- [Background] Weingarten SR, Henning JM, Badamgarav E, Knight K, Hasselblad V, Gano A Jr, Ofman JJ. Interventions used in disease management programmes for patients with chronic illness-which ones work? Meta-analysis of published reports. BMJ. 2002 Oct 26;325(7370):925. doi: 10.1136/bmj.325.7370.925. PMID 12399340